CLINICAL TRIAL: NCT01680432
Title: Effect of the Consumption of a Cheese Enriched With Probiotic Organisms (Bifidobacterium Lactis Bi-07) in Improving Symptoms of Constipation: a Randomized Controlled Trial
Brief Title: Effect of the Consumption of a Cheese Enriched With Probiotic Organisms in Improving Symptoms of Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Univates (Other)
Responsible Party: Principal Investigator, Thaís Rodrigues Moreira, Professor, Centro Universitário Univates
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 033/11
Record Dates: First submitted 2012-08-06; First posted 2012-09-07 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Constipation
Keywords: constipation; probiotics; bifidobacterium; cheese
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic cheese (Experimental): The group received, for 30 days, was instructed to eat 30 g/day of probiotic fresh cheese enriched with Bifidobacterium lactis Bi-07.
  Interventions: Dietary Supplement: Probiotic fresh cheese
- Regular Cheese (Placebo Comparator): The group placebo received, for 30 days, was instructed to consume 30g/day of regular fresh cheese.
  Interventions: Dietary Supplement: Regular Cheese

INTERVENTIONS:
Dietary Supplement: Probiotic fresh cheese — Participants in the intervention group were instructed to drink 30 grams of fresh cheese enriched with probiotics daily for 30 consecutive days.
  Other Names: Fresh cheese enriched with Bifidobacterium lactis Bi-07
  Arms: Probiotic cheese
Dietary Supplement: Regular Cheese
  Arms: Regular Cheese

SUMMARY:
Constipation is a common gastrointestinal motility disorder, chronic condition that often negatively affects the daily lives of patients due to their symptoms, such as infrequent stools, hard stools, straining or painful defecation, cramping, bloating and flatulence. Stress, poor diet and sedentary lifestyle are part of modern lifestyle, which contributes to the onset of constipation. One way to reduce constipation through nutritional management of affected individuals is through consumption of probiotic products, which beneficially affect the development of microbial flora in the intestine, helping to improve the symptoms of constipation. Among these foods, the market is a fresh cheese, plus Bifidobacterium lactis, which according to its maker, when consumed as part of a healthy diet, presents beneficial effects in improving symptoms of constipation.

Hypothesis: The fresh cheese enriched with Bifidobacterium lactis relieves symptoms constipation.

DETAILED DESCRIPTION:
General Objective: To investigate the effect of consumption of fresh cheese enriched with Bifidobacterium lactis in improving symptoms of constipation.

Specific Objectives:

Determine whether the intake of cheese enriched with Bifidobacterium lactis changes:

* frequency of bowel movements;
* straining or pain when defecating;
* format of the faeces;
* sensation of incomplete evacuation;
* sensation of anorectal obstruction and
* use of manual maneuvers to facilitate evacuation.

The food industry is increasingly concerned about produce food that are healthy and able to prevent diseases, in particular, to ensure intestinal health. To verify the effectiveness of these new products on the market is one way to ensure that they have health benefits. Thus, they may be indicated as a treatment for constipation, as part of a healthy lifestyle that includes nutrition and physical activity practice. For this reason, this search is justified.

Type Search:

The research is quantitative, exploratory and experimental. This is a clinical trial randomized and controlled trial.

Population and study sample:

The study population comprised of individuals who will use the Unified Service Health System, the Family Health Strategy,Brazil, participating groups of Nutritional Education. This population is comprised of approximately seventy individuals, but this number is quite relative, it depends on the participation. The approach of research subjects will be done through an invitation, conducted orally through the Community Health Agents (CHA), during home visits monthly. During the period of one month, the CHA invite to attend a lecture given by the student Diane Favretto, who will speak constipation on the subject and propose the participation of stake holders in the research. The stakeholders respond to a questionnaire administered by the student and those who 24 showing symptoms of constipation (according to Rome III criteria), will be part of study, and the sample.

Methodology:

For individuals in the population are classified as constipated, they will responding to a structured questionnaire with closed questions based on criteria Rome III that characterizes the symptoms of constipation. Will be considered constipated individual who has at least two of six symptoms in the questionnaire, 25 at least 25% of the evacuation, in that alternative corresponds to the questionnaire "Often".

Being able to participate in this study, a structured questionnaire, with open and closed questions to assess the lifestyle (dietary habits, intake of net) associated diseases and medications will be made to collect these data.

The weight of the participant will be measured using portable scale brand and the individual is placed standing bare foot in the center of scale with light clothing, with arms out stretched to the side, with out moving. To measure the height measuring tape will be set at flat wall with no baseboard and individuals will be placed in an upright position, standing with bare feet parallel and heels, shoulders and buttocks touching the wall. The Body Mass Index is calculated from data on weight and height (kg / m²) and classified according to the Organization World Health Organization.

Both data will be collected at the neighborhood community hall, where the meetings monthly nutrition education groups are held. Agreeing to participate in the study, the group will receive all necessary instructions and will sign the informed consent. Each participant receives two copies of the word, anda copy shall be given to the student and a copy will be with the participant. Individuals selected to participate in the study will be randomized into two groups: treated group and control group. The treatment group will receive the fresh cheese plus Bifidobacterium lactis Bi-07, with 108 colony forming units per serving. In the placebo group, individuals will receive a fresh cheese, the same brand, with out the addition of probiotics. The products will be packaged or numbered so that neither the researcher nor the participants know what is cheese and what is probiotic cheese placebo. The two groups will be oriented eating a slice of cheese per day (30 grams) for 30 days. This cheese will part of the breakfast. Patients will be advised that, according to the manufacturer's product, both cheeses not present any risk to health. Some patients may not like the taste of cheese. That may be minimized by the use there of in food preparation involving other,as sandwiches and salads, as long as the cheese is not heated, because this way he loses probiotic your property. During this period, all participants will be instructed to continue their normal dietary habits, physical activity and fluid intake. It will also be directed to participants do not make use of other products containing probiotics.

After the intervention period, the questionnaire on the symptoms of constipation is applied again in order to determine whe ther there was a change in bowel habits.

ELIGIBILITY:
Inclusion Criteria:

* adults constipated.

Exclusion Criteria:

* Pregnant women
* Individuals who report to be suffering from other diseases of the intestine;
* Individuals who report not eat cheese, either for reasons of taste or intolerances / food allergies
* Individuals who do not agree to participate and do not sign the term of informed consent

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Increase in frequency of bowel movements after eating probiotic cheese enriched | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Thaís R Moreira, Principal Investigator — University Center Univates
Locations (1):
- Diane Cássia Fravetto, Guaporé, Rio Grande do Sul, Brazil